CLINICAL TRIAL: NCT00937976
Title: Impact of Periodontal Therapy on Metabolic and Inflammatory Markers in Chronic Kidney Disease Patients
Brief Title: Treatment for Periodontal Disease in Dialysis Patients
Acronym: KPU
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: OraPharma (Industry)
Responsible Party: Principal Investigator, Michael Stella, DDS, DDS, University of North Carolina, Chapel Hill
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KPU082008
Record Dates: First submitted 2009-07-09; First posted 2009-07-13 (Estimated); Last update posted 2012-05-07 (Estimated); Status verified 2012-05

CONDITIONS: Periodontal Disease
Keywords: Hemodialysis and peritoneal dialysis
MeSH Terms: conditions — Periodontal Diseases | interventions — Root Planing

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control-delayed periodontal therapy (Other)
  Interventions: Procedure: Periodontal Scaling and Root Planing
- Intensive Periodontal Therapy (Other)
  Interventions: Procedure: Periodontal Scaling and Root Planing

INTERVENTIONS:
Procedure: Periodontal Scaling and Root Planing — Participants will take antibiotics prior to dental treatment. Periodontal treatment or a deep cleaning (with local anesthesia or numbing) will be performed to remove plaque and tartar around the teeth and gums. A small amount of antibiotics (minocycline) will be placed around the gums to help fight bacteria and inflammation.

SUMMARY:
The primary objective is to test the hypothesis that periodontal intervention in dialysis patients who have both periodontal disease and a historically high burden of cardiovascular disease will result in a reduction of inflammatory markers and improvement markers of nutrition health like albumin. Patients will be randomized to one of two treatment arms: intensive periodontal therapy or control-delayed periodontal therapy. Eligible patients will have 5 study visits over 7 to 12 months.

DETAILED DESCRIPTION:
The burden of cardiovascular disease (CVD) is well known to those taking care of patients with chronic kidney disease (CKD). Myocardial infarction, sudden death, or stroke, remain leading causes of death and disability, especially for those patients receiving dialysis therapy (Foley 2003). Traditional risk factors (Wilson, D'Agostino et al. 1998) only partially explain the burden of CVD (Longenecker, Coresh et al. 2002).

Our research team has been studying the potential role of periodontal disease in explaining the excess burden of CVD in the CKD population. Periodontitis is an inflammatory disease caused by an infection of predominately gram negative organisms (Pihlstrom, Michalowicz et al. 2005) and has been well-studied in other populations as a CVD risk factor (DeStefano, Anda et al. 1993; Mattila, Valtonen et al. 1995; Beck, Garcia et al. 1996; Joshipura, Rimm et al. 1996; Morrison, Ellison et al. 1999; Hujoel, Drangsholt et al. 2000; Wu, Trevisan et al. 2000; Howell, Ridker et al. 2001; Hujoel, Drangsholt et al. 2001; Hung, Willett et al. 2003; Joshipura, Hung et al. 2003; Tuominen, Reunanen et al. 2003; Hung, Joshipura et al. 2004; Pussinen, Alfthan et al. 2004; Pussinen, Nyyssonen et al. 2005; Saremi, Nelson et al. 2005). It has also been demonstrated to accelerate preclinical and clinical atherosclerosis (Loesche, Schork et al. 1998; Arbes, Slade et al. 1999; Genco 1999). In an observational cohort of 168 patients receiving maintenance hemodialysis followed for 18 months, severe and moderate periodontitis was strongly associated with death of cardiovascular causes independent of traditional risk factors (unpublished data). A very high prevalence of periodontal disease in patients with various stages of CKD has been observed. In this population, periodontal disease was associated with a low serum albumin and malnutrition (Kshirsagar, Craig et al. 2007).

We present a randomized interventional small exploratory study to assess study feasibility and to determine whether the treatment of periodontal disease in maintenance dialysis patients reduces markers of inflammation and improves markers of nutrition. The existent data support an intervention trial, rather than additional observational studies. There are a multitude of epidemiological studies, including our studies, which confirm an association of periodontal disease and cardiovascular disease (DeStefano, Anda et al. 1993; Mattila, Valtonen et al. 1995; Beck, Garcia et al. 1996; Joshipura, Rimm et al. 1996; Morrison, Ellison et al. 1999; Hujoel, Drangsholt et al. 2000; Wu, Trevisan et al. 2000; Howell, Ridker et al. 2001; Hujoel, Drangsholt et al. 2001; Hung, Willett et al. 2003; Joshipura, Hung et al. 2003; Tuominen, Reunanen et al. 2003; Hung, Joshipura et al. 2004; Pussinen, Alfthan et al. 2004; Pussinen, Nyyssonen et al. 2005; Saremi, Nelson et al. 2005). Thus, the time is right for conducting a hypothesis-driven intervention trial.

ELIGIBILITY:
Inclusion Criteria:

* Presence of 12 or more teeth
* Presence of moderate to severe periodontal disease (2 or more teeth with at least 6 mm Clinical Attachment Loss and at least 1 site with Probing Depth > 5 mm)
* Receiving dialysis for at least 3 months
* English speaking
* Ability and willingness to give written informed consent for participation in the study
* Age 18 to 80 years
* Twelve or more teeth

Exclusion Criteria:

* Any severe co-morbid conditions likely to affect life expectancy within 1 year (for example, metastatic cancer)
* Any condition that would, in the judgement of the clinician, be a contraindication to dental treatment
* Dementia
* Pregnancy or lactation
* Inability to take oral medications
* Allergy or intolerance to minocycline, tetracyclines or polygycolate polymers
* Allergy to both penicillin and clindamycin
* Severe dental caries, pulpal or mucosal disease that would interfere with periodontal therapy
* Inability or unwillingness to follow the study protocol

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2008-08; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
Serum Albumin, IL-6, CRP | 6 months

SECONDARY OUTCOMES:
HbA1c, periodontal probing | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Steven Offenbacher, DDS, PhD, Principal Investigator — UNC Chapel Hill
Locations (1):
- GO Health Center, School of Dentistry, University of North Carolina-Chapel Hill, Chapel Hill, North Carolina, United States

REFERENCES:
- [Derived] Wehmeyer MM, Kshirsagar AV, Barros SP, Beck JD, Moss KL, Preisser JS, Offenbacher S. A randomized controlled trial of intensive periodontal therapy on metabolic and inflammatory markers in patients With ESRD: results of an exploratory study. Am J Kidney Dis. 2013 Mar;61(3):450-8. doi: 10.1053/j.ajkd.2012.10.021. Epub 2012 Dec 20. PMID 23261122